CLINICAL TRIAL: NCT03254992
Title: Motor Learning Transfer Between Real and Virtual Environments in Autism Spectrum Disorder.
Brief Title: Real and Virtual Environments in Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carlos Bandeira de Mello Monteiro, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 55498016.1.0000.5390
Record Dates: First submitted 2017-06-01; First posted 2017-08-21 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ASD - Abstract task (Experimental): Experimental group using Kinect with more virtual activity.
  Interventions: Device: ASD - Abstract task
- ASD - Tangible task (Experimental): Experimental group using Keyboard with more real activity.
  Interventions: Device: ASD - Tangible task
- TD - Abstract task (Active Comparator): Control group using Kinect with more virtual activity.
  Interventions: Device: TD - Abstract task
- TD - Tangible task (Active Comparator): Control group using Keyboard with more real activity.
  Interventions: Device: TD - Tangible task

INTERVENTIONS:
Device: ASD - Abstract task — Experimental group using Kinect with more virtual activity.
  Arms: ASD - Abstract task
Device: ASD - Tangible task — Experimental group using Keyboard with more real activity.
  Arms: ASD - Tangible task
Device: TD - Abstract task — Control group using Kinect with more virtual activity.
  Arms: TD - Abstract task
Device: TD - Tangible task — Control group using Keyboard with more real activity.
  Arms: TD - Tangible task

SUMMARY:
Individuals with Autism Spectrum Disorder (ASD) are known to have difficulty with socio-communicative functioning and restricted or repetitive behaviors or interests, and there is considerable evidence that the majority also struggle with associated emotional problems. Speech is typically delayed or may regress, comprehension is impaired, if not at the word level, then at the level of sentences, nonverbal and verbal language are affected, and pretend play is delayed or absent, some children are nonverbal or have sparse, impoverished, poorly articulated, and grammatical speech. Objective: To assess in which interface has ASD best performance or functionality. Method: Will be evaluated 100 individuals divided into two groups: 50 individuals with diagnosis of Autistic Spectrum Disorder (ASD-group), aged 7 to 15 years old, males and females; and 50 individuals with typical development (TD-group) matched by age and sex to the ASD-group. Individuals with comorbidities and functional disabilities that would impede the completion of the task were excluded.

DETAILED DESCRIPTION:
Will be evaluated 100 individuals divided into two groups: 50 individuals with diagnosis of Autistic Spectrum Disorder (ASD-group), aged 7 to 15 years old, males and females; and 50 individuals with typical development (TD-group) matched by age and sex to the ASD-group. The ASD-group will be recruited from GAPI - Special Education in São Bernardo do Campo, São Paulo, Brazil, which is a school for children and adolescents with pervasive developmental disorders.

For a diagnosis of ASD, apart from qualitative alterations in social communication and interaction (criterion A) in addition to stereotyped, repetitive, restricted behavior patterns (criterion B), that present in the early developmental period (criterion C), it is also required that these "symptoms cause clinically significant impairment in social, occupational and other important areas of current functioning" (criterion D), and that they are not better explained otherwise (criterion E). Given this information these items will be taken into consideration and the group was well evaluated.

With the purpose to homogenize the sample, will be only included ASD with the 1st level to 5th education to grade elementary.

Instrument For data collection will be used a gaming software created in partnership with the Information Systems group of School of Arts, Sciences and Humanities, EACH-USP.

The game offers task of "Timing" Coincident, which when executed are displayed on the computer screen 10 balls accessing (red light) in sequence until the last ball, which is considered the target (green light). The participant can have immediate feedback of hit or task error by different sounds (Auditory Interaction) and through visual images (Visual Interaction) that change colors, that will be previously shown to him.

Task Coincident Timing In the more tangible button-press task, the individuals will be required to 'intercept' a falling virtual object at the moment it reached the interception point by pressing a button on the computer's keyboard. In the more abstract, less tangible task, they were instructed to 'intercept' the virtual object by making a hand movement (i.e., a waving gesture) in a virtual environment.

The magnitude and direction of each participant's error in anticipating the light's "arrival" at the end of the runway, in milliseconds, is recorded by the game.

Objective the game is to evaluate the difference in time between the participant's execution of the response and the arrival of the object at the target location, overall temporal accuracy, and hence coincidence-anticipation timing skill.

The software provides a "user login" for each research participant, where the following data are stored: Participant name; Date of birth; sex; Pathology type; Researcher name.

Procedures The participants will be positioned comfortably in a chair adjusted according to size and needs along with a footrest so that they will be positioned properly to enable task execution. Before starting the task, the operation of the game will be verbally explained and a demonstration will be offered by the examiner. Runtime will be noted in each experimental stage, as explained below: acquisition (A), retention (R), and transfer (T).

All participants made 20 trial acquisitions, 5 retention trials after 5 minutes with no contact with the task and 5 transfer trials immediately after retention trials. Thus, each participant will have 30 trials. During acquisition and retention trials, the bubbles simulate a dropped light movement with 0.5 seconds between each bubble and 5 seconds between the first and last bubble.

The subjects will perform alternating interfaces for the same task, Kinect for Windows (gesture task with virtual environments), Keyboard (button press with tangible environments), and both groups will carry out the transfer phase on Touch Screen interface. The subjects of each group (ASD and TD) will be divided into 2 groups, group A and group B, according to the order of interfaces to carry out the task; Group A will perform the abstract task (kinect with more virtual activity) and then the tangible task (keyboard with more real activity), and the group B, will perform the reverse process.

ELIGIBILITY:
Inclusion Criteria:

* need to understand the task, assessed by the ability to properly perform three attempts explanatory statement by the evaluator.

Exclusion Criteria:

* of incomprehension.
* no completion of the task.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2016-11-02 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Change in performance, measured by coincident timing task | 1 day
  The participants who will perform the abstract task first, will present decrease on performance, measured by the coincident timing task.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos BM Monteiro, Ph.D., Principal Investigator — University of Sao Paulo
Locations (1):
- Escola de Artes,Ciencias e Humanidades da Universidade d Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided